CLINICAL TRIAL: NCT04168528
Title: Phase I/IIa Study to Evaluate the Safety, Biodistribution, Radiation Dosimetry and Tumor Imaging Potential of 68GaNOTA-Anti-MMR-VHH2, a New Radiopharmaceutical for in Vivo Imaging of Tumour-Associated Macrophages by Means of PET : UZBRU_VHH2_1
Brief Title: Phase I/IIa Study of 68GaNOTA-Anti-MMR-VHH2 for PET/CT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: UZBRU_VHH2_1; 2017-001471-23 (EudraCT Number)
Record Dates: First submitted 2019-11-07; First posted 2019-11-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Malignant Solid Tumor; Breast Cancer; Melanoma (Skin)
Keywords: PET/CT; MMR-PET/CT; Macrophage PET/CT
MeSH Terms: conditions — Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part I: safety, tolerability, biodistribution and dosimetry (Experimental): Phase I
  Interventions: Drug: 68GaNOTA-Anti-MMR-VHH2
- Part II: tumor targeting potential and correlation to IHC (Experimental): Phase II
  Interventions: Drug: 68GaNOTA-Anti-MMR-VHH2

INTERVENTIONS:
Drug: 68GaNOTA-Anti-MMR-VHH2 — Injection of the radiopharmaceutical and PET/CT imaging

SUMMARY:
Phase I study to evaluate the human safety and tolerability, biodistribution and dosimetry of 68GaNOTA-Anti-MMR-VHH2

Phase IIa study to evaluate tumour uptake of 68Ga-NOTA-anti-MMR-VHH2 in patients with breast cancer or melanoma. To correlate uptake of 68Ga-NOTA-anti-MMR-VHH2 in cancer lesions to immunohistological MMR staining after resection or biopsy of the same lesion.

ELIGIBILITY:
PART I:

Inclusion Criteria:

Patients will only be included in the study if they meet all of the following criteria:

* Patients who have given informed consent
* Patients at least 18 years old
* Patients with local, locally advanced or metastatic disease of a malignant solid tumor. In order to minimize partial volume effect the diameter of at least 1 tumor lesion should be ≥ 10 mm in short axis for invaded adenopathies and ≥ 10 mm in long axis for all other types of lesions.

Exclusion Criteria:

Patients will not be included in the study if one of the following criteria applies:

* Eastern Cooperative Oncology Group (ECOG) performance status 3 or higher
* Pregnant patients
* Breast feeding patients
* Patients with abnormal liver (Bilirubin ≥1.5 x ULN, ALT (SGPT) ≥3 x ULN) or kidney function (Serum creatinine clearance ≤50 ml/min as calculated with Cockcroft-Gault formula)
* Patients with recent (< 1 week) gastrointestinal disorders (CTCAE v4.0 grade 3 or 4) with diarrhea as major symptom
* Patients with any serious active infection
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test radiopharmaceutical
* Patients who cannot communicate reliably with the investigator
* Patients who are unlikely to cooperate with the requirements of the study
* Patients who are unwilling and/or unable to give informed consent
* Patients at increased risk of death from a pre-existing concurrent illness
* Patients who participated already in this study

PART II:

Inclusion Criteria:

Patients will only be included in the study if they meet all of the following criteria:

* Patients who have given informed consent
* Patients at least 18 years old
* Patients diagnosed with a local, locally advanced or metastatic disease, with any of the following cancer types :
* Triple-negative breast carcinoma,
* Hormone-receptor negative (HR-), HER2+ breast carcinoma, with HER2-expression defined as HER2+ on ISH or 3+ on IHC, as determined by local assessment on any of the available cancer tissues
* Melanoma
* Patients who have had a biopsy of at least one lesion or who are planned to undergo standard-of-care resection or biopsy of at least one lesion, in order to minimize partial volume effect, the diameter of that lesion should be ≥ 10 mm in short axis for invaded adenopathies and ≥ 10 mm in long axis for all other types of lesions.

Exclusion Criteria:

Patients will not be included in the study if one of the following criteria applies:

* Eastern Cooperative Oncology Group (ECOG) performance status 3 or higher
* Pregnant patients
* Breast feeding patients
* Patients with recent (< 1 week) gastrointestinal disorders (CTCAE v4.0 grade 3 or 4) with diarrhea as major symptom
* Patients with any serious active infection
* Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the test radiopharmaceutical
* Patients who cannot communicate reliably with the investigator
* Patients who are unlikely to cooperate with the requirements of the study
* Patients who are unwilling and/or unable to give informed consent
* Patients at increased risk of death from a pre-existing concurrent illness
* Patients who participated already in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety of 68GaNOTA-Anti-MMR-VHH2: reported as type, frequency and severity (graded according to the CTCAEv5) (Part I). | Before injection up until 6 hrs after injection
  Assessed using physical examination and blood sampling for hematology and clinical chemistry.
Human biodistribution using blood sampling and PET/CT imaging: reported as relative uptake values per organ at 10, 90 and 150 minutes per individual subject and as a mean over all subjects (Part I). | Immediately after injection up to 3 hrs after injection
  Measured in standard uptake values in PET/CT imaging and expressed in relation to the injected activity.
Human dosimetry using PET/CT imaging data: radiation dose to individual organs and the equivalent dose for the whole body of each subject and as a mean over all subjects (Part I). | 10 min up to 3 hrs after injection
  Dosimetry will be calculated using the OLINDA software.
Tumor targeting potential using PET/CT and correlation to immunohistological MMR staining after resection: assessed using correlation coefficient (Part II). | Resection of lesion up to 14 days after PET/CT
  PET/CT and immunohistochemistry will be assessed using a semi-quantitative scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tony LAHOUTTE, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Uz Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No